CLINICAL TRIAL: NCT00294099
Title: A Phase I-II, Randomized, Controlled, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine Given Alone or With Aluminum Hydroxide to Healthy Elderly Adults
Brief Title: H5 Vaccine Alone or With Aluminum Hydroxide in Elderly Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0141
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
Keywords: A/H5N1, Influenza, Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 2 (Experimental): 120 subjects to receive 45 mcg of inactivated influenza A/H5N1 vaccine without aluminum hydroxide.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 3 (Experimental): 60 subjects to receive 15 mcg of inactivated influenza A/H5N1 vaccine with aluminum hydroxide.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 4 (Experimental): 60 subjects to receive 15 mcg of inactivated influenza A/H5N1 vaccine without aluminum hydroxide.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 8 (Experimental): 60 subjects to receive 3.75 mcg of inactivated influenza A/H5N1 vaccine without aluminum hydroxide.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 7 (Experimental): 60 subjects to receive 3.75 mcg of inactivated influenza A/H5N1 vaccine with aluminum hydroxide.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 1 (Experimental): 120 subjects to receive 45 mcg of inactivated influenza A/H5N1 vaccine with aluminum hydroxide.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 5 (Experimental): 60 subjects to receive 7.5 mcg of inactivated influenza A/H5N1 vaccine with aluminum hydroxide.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 6 (Experimental): 60 subjects to receive 7.5 mcg of inactivated influenza A/H5N1 vaccine without aluminum hydroxide.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)

INTERVENTIONS:
Biological: Aluminum hydroxide — Aluminum hydroxide adjuvant.
  Arms: 1; 3; 5; 7
Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur) — Inactivated monovalent subvirion influenza H5N1 vaccine. Supplied in 0.5 mL unit dose vials as a sterile solution for IM injection. Dosages: 45 mcg, 15 mcg, 7.5, mcg, or 3.75 mcg administered with or without aluminum hydroxide adjuvant on Days 0 and 28.

SUMMARY:
The purpose of this study is to compare how the body reacts to different strengths of the new A/H5N1 flu vaccine when given with the addition of aluminum hydroxide adjuvant and provide dosing information. How the body's immune system responds to the new H5N1vaccine with aluminum hydroxide approximately 1 month following receipt of 2 doses of vaccine will also be evaluated. The vaccine is given as an injection or shot in the arm. Volunteer participants in this study will be 600 healthy elderly adults, aged 65 years and older. Participants will be randomly assigned to 4 different dosage groups of vaccine, either with or without adjuvant, for a total of 8 different groups. Volunteers will participate in the study for 7 months. Each individual will receive two vaccinations, the second 28 days after the first. In addition to visits for these vaccinations, subjects will return to the clinic for physical evaluations and blood sample collection 6 times during the course of this study.

DETAILED DESCRIPTION:
This is a double-blind, randomized, controlled, dose-ranging, Phase I-II study in healthy ambulatory elderly adults. The primary objectives are to: determine the dose-related safety of subvirion-inactivated H5N1 vaccine adjuvanted with aluminum hydroxide in healthy elderly adults (65 years of age and older); determine the potential for aluminum hydroxide to enhance the immune response to subvirion inactivated H5N1 vaccine in healthy elderly adults approximately 1 month following receipt of 2 doses of vaccine; and provide information for the selection of the best dosage level for further studies. A secondary objective is to evaluate dose-related immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination. Approximately 600 elderly subjects are planned for enrollment. Subjects will be screened for health status by history and targeted physical examination. Subjects who meet the entry criteria for the study will be randomized into 8 groups to receive 2 doses of nonadjuvanted or aluminum hydroxide-adjuvanted influenza A/H5N1 vaccine containing 3.75, 7.5, 15, or 45 micrograms of hemagglutinin (HA) by intramuscular injection. The first vaccination will occur on Day 0. Symptoms and signs will be assessed in the clinic for at least 15 minutes after inoculation, and subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 7 days after each immunization. Subjects will be encouraged to take their temperature around the same time each day. All subjects will return to the clinic on Days 2 and 8 after each vaccination for assessment of AEs and concomitant medications, as well as a targeted physical examination if indicated. Memory aids will be reviewed at each visit. At approximately Day 28 after the first vaccination, subjects will return to the clinic for blood sample collection and safety follow-up, followed by a second vaccination. Safety follow-up will be identical to that performed after the first vaccination. Approximately 56 days after first immunization (or about 28 days after the second vaccination), subjects will return to the clinic for immunogenicity blood sample collection, AE and concomitant medication assessments, and targeted physical examinations (if indicated). At approximately Day 208 (7 months after the first vaccination), subjects will return to the clinic for a final immunogenicity blood sample collection and for follow-up, which includes a targeted physical examination if indicated. The duration of the study treatment for each subject will be about 7 months. The primary study endpoints include: AE or serious adverse event (SAE) information; proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 1:40 against influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine; proportion of subjects in each dose group achieving a serum hemagglutination inhibition (HAI) antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine; geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 28 days after receipt of the second dose of vaccine; and GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 28 days after receipt of the second dose of vaccine. The secondary endpoints include: GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; GMT and frequency of 4-fold or greater increases i

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory adults aged 65 and older
* Are in good health, as determined by vital signs (heart rate less than 100 bpm, blood pressure [systolic less than or equal to 160 mm Hg and diastolic less than or equal to 90 mm Hg] oral temperature less than 100.0°F), medical history to ensure stable medical condition, and targeted physical examination based on medical history
* Are able to understand and comply with planned study procedures
* Provide written informed consent prior to initiation of any study procedures

Stable medical condition - no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal, aluminum hydroxide, and chicken protein).
* Have immunosuppression as a result of an underlying illness or treatment, or used anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Have any malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder diagnosed or treated actively during the past 5 years.
* Have long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids ( > 800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate.) Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long there has been no dose adjustment within the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Heart Association Functional Class III or IV); an arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack).
* Have a history of severe reactions following immunization with influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week prior to vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 7- to 8-month study period.
* Have any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (but does not exclude documented placebo recipients).
* Have a known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Planned to travel outside of the USA in the time between the first vaccination and 56 days following the first vaccination.
* Have any diagnosis of dementia or associated concomitant medications (e.g., Aricept) used for treating dementia.
* Have a history of Guillain Barre syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 28 days after receipt of the second dose of vaccine. | Approximately day 56.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 28 days after receipt of the second dose of vaccine. | Approximately day 56.
Proportion of subjects in each dose group achieving a serum hemagglutination inhibition (HAI) antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine. | Approximately day 56.
Proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine. | Approximately day 56.
Adverse event (AE) or serious adverse event (SAE) information (solicited in the clinic and via memory aids, concomitant medications, and periodic targeted physical assessment). | Adverse events will be collected through 28 days following the 2nd dose of vaccine (day 56). Serious adverse events will be collected throughout the study through day 208.

SECONDARY OUTCOMES:
Development of serum antibody responses against antigenically drifted variants of H5N1 influenza virus. | Day 0, and at days 28, 56, and 208 after the first immunization.
GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine. | Day 0, and at days 28, 56, and 208 after the first immunization.
GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine. | Day 0, and at days 28, 56, and 208 after the first immunization.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Brady RC, Treanor JJ, Atmar RL, Keitel WA, Edelman R, Chen WH, Winokur P, Belshe R, Graham IL, Noah DL, Guo K, Hill H. Safety and immunogenicity of a subvirion inactivated influenza A/H5N1 vaccine with or without aluminum hydroxide among healthy elderly adults. Vaccine. 2009 Aug 13;27(37):5091-5. doi: 10.1016/j.vaccine.2009.06.057. Epub 2009 Jul 3. PMID 19577636